CLINICAL TRIAL: NCT00554190
Title: A Prospective, Multi-Center, Randomized, Controlled, Subject-Blinded Study to Evaluate the Safety and Effectiveness of AdvaCoat Sinus Gel Following Endoscopic Ethmoid Sinus Surgery
Brief Title: Study to Evaluate Safety and Effectiveness of AdvaCoat Sinus Gel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carbylan Therapeutics, Inc. (Industry)
Responsible Party: Marcee Maroney, V.P. Marketing and Clinical Affairs, Carbylan BioSurgery, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACOT 1.0
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Results first posted 2009-04-23 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-03

CONDITIONS: Ethmoid Sinusitis; Rhinosinusitis
Keywords: rhinosinusitis, ethmoid
MeSH Terms: conditions — Ethmoid Sinusitis; Rhinosinusitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AdvaCoat compared to Merogel Injectable Bioresorbable Nasal Dressing
  Interventions: Device: AdvaCoat sinus gel
- 2 (Active Comparator): Merogel Injectable Bioresorbable Nasal Dressing compared to AdvaCoat
  Interventions: Device: Merogel Injectable

INTERVENTIONS:
Device: AdvaCoat sinus gel — A sterile,viscoelastic, bioresorbable gel composed of highly purified hyaluronan, a naturally occurring constituent of tissues in the body
  Arms: 1
Device: Merogel Injectable — Bioresorbable hyaluronic acid product
  Other Names: Merogel
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of AdvaCoat® sinus gel, a nasal/sinus dressing, for adhesion prevention following endoscopic ethmoid sinus surgery. Subjects were randomized to receive AdvaCoat applied to the right or left middle meatus tissues and Merogel applied to the middle meatus tissues on the opposite side.

DETAILED DESCRIPTION:
Chronic rhinosinusitis is a very common condition, affecting 35 million Americans each year. All paranasal sinuses need ventilation to prevent infection and inflammation. Sinus ventilation occurs through the ostia into the nose. When rhinosinusitis occurs, the mucous membranes of the sinuses become swollen, resulting in ostia closure. Functional endoscopic sinus surgery (FESS) is a minimally invasive surgical procedure that opens the sinus ostia.

The most common unwanted side effect of the FESS procedure is the formation of adhesions (fibrous bands) in the area of surgery. These bands (adhesions) can prevent proper ventilation and drainage from the paranasal sinuses.

Various hyaluronan based biomaterials are now available and in common use to provide a post-surgical nasal dressing which is absorbable, can prevent adhesion formation, and eliminate the pain and tissue abrasion caused by removal of non-absorbable nasal packing.

AdvaCoat is a bioresorbable hyaluronan gel that conforms to mucosal surfaces and provides a post-surgical nasal dressing to prevent adhesion formation as tissues heal.

ELIGIBILITY:
Inclusion Criteria:

Patients who:

1. Have bilateral chronic rhinosinusitis confirmed by physical exam, clinical history, and prior radiography
2. Have bilateral ethmoid sinus disease
3. Are scheduled for bilateral anterior or total ethmoidectomy

Exclusion Criteria:

1. Unilateral ethmoid sinus disease
2. Partial resection of middle turbinates, unilateral or bilateral

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew N. Goldberg, MD, Principal Investigator — University of California, San Francisco, Medical Center
Locations (4):
- United States (4):
  - Alabama Nasal & Sinus Center, Birmingham, Alabama
  - University of California, San Francisco, Dept of Otolaryngology, San Francisco, California
  - Northwestern University Medical Center, Department of Otolaryngology, Chicago, Illinois
  - Cleveland Nasal Sinus & Sleep, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject treatment: May 2007. Last subject treatment: December 2007.
Pre-assignment Details: A total of 29 subjects were treated. Nineteen subjects were followed through 60 days post-treatment.
Groups:
- AdvaCoat and Merogel: AdvaCoat compared to Merogel Injectable. Subjects were randomized to receive AdvaCoat applied to the right or left middle meatus tissues and Merogel applied to the middle meatus tissues on the opposite side.
Period: Overall Study
Arm/Group | AdvaCoat and Merogel
Started | 29 (29 subjects treated.)
Completed | 19 (10 subjects did not complete the Termination Study Forms)
Not Completed | 10
Not completed — Termination forms not completed | 10

BASELINE CHARACTERISTICS:
Groups:
- AdvaCoat and Merogel Injectable: AdvaCoat compared with Merogel Injectable
Arm/Group | AdvaCoat and Merogel Injectable
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adhesion as Measured by the Synechia (Adhesion) Scale
Description: Synechia (adhesion) scale range of 0 = No visible synechia to 3 = Complete scarring between the middle turbinate and lateral nasal wall was used in the assessment.
Time Frame: Post-operative through 60 days
Population: There were 19 participants that completed the final follow-up visit at 60 days.
Measure: Number; unit: Participants
Groups:
- Merogel Injectable: Merogel Injectable compared to AdvaCoat
- AdvaCoat Sinus Gel: AdvaCoat compared to MeroGel Injectable
Arm/Group | Merogel Injectable | AdvaCoat Sinus Gel
Number analyzed (Participants) | 19 | 19
Participants
  0 (no visible synechia) | 14 | 13
  1 (one or several visible synechia) | 4 | 5
  2 (synechia w/ interference to sinus ventilation ) | 1 | 1
  3 (complete scarring) | 0 | 0

2. Primary Outcome: Number of Participants With Solicited and Recorded Adverse Events
Description: All reported events were coded to a standard set of terms using the MedDRA adverse event dictionary. Adverse events were listed and summarized.
Time Frame: Post-operative through 60 days
Population: There were 19 participants who completed the 60 day follow up visits for analysis.
Measure: Number; unit: Participants
Arm/Group | Merogel Injectable | AdvaCoat Sinus Gel
Number analyzed (Participants) | 19 | 19
Participants
  Mucopurulent drainage | 1 | 2
  Mucopurulent drainage with polypoid swelling | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No